CLINICAL TRIAL: NCT06385808
Title: Efficacy and Safety of Mitoxantrone Hydrochloride Liposome Combined With Thiotepa, Busulfan and Fludarabine Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Efficacy and Safety of MTBF Conditioning Regimen for Salvageable Allo-HSCT in the Treatment of R/R AML
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2023-XK014
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Relapse Leukemia; Refractory Acute Myeloid Leukemia; Conditioning; Hematopoietic Stem Cell Transplantation
Keywords: relapsed or refractory acute myeloid leukemia; conditioning regimen; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Thiotepa; Busulfan; fludarabine

STUDY DESIGN:
Intervention Model Description: The relapsed or refractory acute myeloid leukemia patients will pretreated with the MTBF regimen prior to salvageable allogeneic hematopoietic stem cells. The one-year recurrence-free survival after transplantation of these patients and the safty of the MTBF regimen will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MTBF regimen group (Experimental): The relapsed or refractory acute myeloid leukemia patients will pretreated with the MTBF regimen prior to salvageable allogeneic hematopoietic stem cells.
  Interventions: Drug: MTBF regimen

INTERVENTIONS:
Drug: MTBF regimen — The subjects will be treated with mitoxantrone hydrochloride liposome combined with thiotepa, busulfan and fludarabine as conditioning regimen prior to allo-HSCT.
  Mitoxantrone hydrochloride liposome 24mg/m^2 ivgtt d-7; Ctepide 5mg/kg ivgtt d-6~-5; Busulfan 0.8mg/kg q6h ivgtt d-4~-2; Fludarabine 50mg/m^2 ivgtt d-4~-2.
  Other Names: Mitoxantrone Hydrochloride Liposome; Thiotepa; Busulfan; Fludarabine

SUMMARY:
The primary objective of this study was to evaluate the efficacy of MTBF conditioning regimen of salvageable allo-HSCT in patients with relapsed or refractory acute myeloid leukemia. The secondary purpose of the study was to observe the safety of MTBF regimen in these patients.

DETAILED DESCRIPTION:
High-intensity conditioning regimen prior to allogeneic hematopoietic stem cell transplantation (allo-HSCT) can maximize the clearance of leukemia cells, but is often associated with increased pretreatment-related toxicity and transplant-related mortality. In order to enhance its anti-tumor effect without increasing or even decreasing its tissue toxicity, and then prolong the overall survival of AML patients, we optimized the conditioning regimen before allo-HSCT transplantation: (1) The classical Thiotepa/Busulfan/Fludarabine (TBF) regimen will be adopted to reduce the conditioning associated toxicity, ensure graft implantation to the maximum extent and reduce the recurrence rate; ② At the same time, mitoxantrone hydrochloride liposome will be added to avoid the disadvantages of weak immunosuppressive effect and weak anti-leukemia effect, and MTBF pretreatment scheme will be finally explored. It has been applied in the pre-treatment of salvage allo-HSCT in 3 patients with relapsed and refractory acute myeloid leukemia with good safety. Up to the present follow-up time of 4 months, all 3 patients have disease free survival. To evaluate the safety and efficacy of this protocol, we intend to include more patients undergoing salvage allo-HSCT for relapsed or refractory (R/R) AML.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with the follow-up;
* Age 18-65 years old (including upper and lower limits);
* No gender limitation
* Relapsed or refractory (R/R) acute myeloid leukemia can not achieve complete remission by chemotherapy, and has the indication of salvage allogeneic hematopoietic stem cell transplantation.
* R/R AML was defined as: ① Initial treatment cases that failed after 2 courses of standard chemotherapy; ② After CR consolidation and intensive treatment, relapse within 12 months; ③ Recurred 12 months later, but conventional chemotherapy was ineffective; ④ Two or more relapses; ⑤ Extramedullary leukemia persists; ⑥Leukemia cells in peripheral blood or the proportion of bone marrow original cells >0.050 or the occurrence of extramedullary leukemia cell infiltration after CR.
* Could tolerate allogeneic hematopoietic stem cell transplantation.

Exclusion Criteria:

* Hypersensitivity to any investigational drug or its components;
* Uncontrolled systemic diseases (e.g. active infections, uncontrolled hypertension, diabetes, etc.)
* Cardiac function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval>480 ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Serious and uncontrolled arrhythmia requiring drug treatment;
  4. American New York Heart Association rating ≥ III degree;
  5. Cardiac ejection fraction (LVEF) is less than 60%;
  6. History of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or He has any arrhythmia requiring treatment, clinical history of serious pericardial disease, or acute ischemia or activity ECG evidence of abnormal conduction system;
* Active infection of hepatitis B and hepatitis C;
* Human immunodeficiency virus (HIV) infection;
* Patients with other malignant tumors;
* History of drug abuse (non-medical use of narcotic drugs or psychotropic drugs) or history of drug dependence (sedative hypnotics, analgesics, narcotics, stimulants and psychotropic drugs, etc.);
* History of mental illness or cognitive impairment;
* Other investigators determined that participation in this study was not appropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years post transplantation
  Disease activity in patients after transplantation

SECONDARY OUTCOMES:
Incidence and Severity of non-hematological adverse events (NCI CTCAE v5.0) | from the beginning of the conditioning regimen to 2 years post transplantation
  The incidence and severity of non-hematological adverse events were evaluated using NCI CTCAE v5.0 criteria.
Neutrophil recovery time | 1 month post transplantation
  Peripheral blood neutrophil count (ANC) ≥0.5×10^9/L for three consecutive days without blood transfusion support
Platelet recovery time | 1 month post transplantation
  Peripheral blood platelet (PLT) ≥20×10^9/L for three consecutive days without blood transfusion support.
OS | From date of diagnosis until the end of follow-up or the date of death from any couse. Time rage: 6 months post transplantation, 12 months post transplantation.
  Overall survival
PFS | From date of diagnosis until the end of follow-up or disease progression. Time rage: 6 months post transplantation, 12 months post transplantation.
  Progression-free survival

OTHER OUTCOMES:
aGVHD | At day 100 post transplantation
  The incidence of acute graft versus host disease

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Wang, M.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University